CLINICAL TRIAL: NCT02087475
Title: Randomized Open-label Phase III Study Comparing Perioperative FOLFIRI Versus Adjuvant FOLFIRI in Resectable Advanced Colorectal Cancer Failed to Oxaliplatin-containing Treatment
Brief Title: Perioperative FOLFIRI VS Adjuvant FOLFIRI in Resectable Advanced CRC Failed to Oxaliplatin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ping Lan, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAH 5010 CRC
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Neoplasms; Effects of Chemotherapy; Surgery; Metastasis; Local Neoplasm Recurrence
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasm Recurrence, Local | interventions — Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant therapy arm (Experimental): FOLFIRI * 6 cycles +/- radiotherapy -> surgery -> FOLFIRI * 6 cycles
  Interventions: Drug: Irinotecan; Drug: 5-fluorouracil; Radiation: Local radiotherapy; Procedure: R0 resection
- Adjuvant therapy arm (Active Comparator): Surgery -> FOLFIRI * 12 cycles +/- radiotherapy
  Interventions: Drug: Irinotecan; Drug: 5-fluorouracil; Radiation: Local radiotherapy; Procedure: R0 resection

INTERVENTIONS:
Drug: Irinotecan
Drug: 5-fluorouracil
Radiation: Local radiotherapy
Procedure: R0 resection

SUMMARY:
Colorectal cancer (CRC) is one of the most leading causes of cancer death in China. Although multiple treatment modalities including surgery, radiotherapy and chemotherapy have been developed, the prognosis of advanced CRC still remains poor. While around 30% of resectable advanced CRC could be cured. This study is designed to compare perioperative FOLFIRI versus adjuvant FOLFIRI in resectable advanced CRC who exposed to oxaliplatin in open-label, phase III mode.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-80
* ECOG score: 0 or 1
* Histological confirmed of Colorectal Adenocarcinoma
* History of exposure to oxaliplatin
* With local recurrent or metastatic focus
* Tumor resectable confirmed by at less 3 hepatobiliary surgeon
* Informed content acquired

Exclusion Criteria:

* History of Exposure to Irinotecan
* Received surgery in recently 4 weeks or did not recover from surgery
* Other history of cancer in recent 5 years
* Fluorouracil allergy or dihydropyrimidine dehydrogenase defect
* Women with potential pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2011-01; Primary Completion 2021-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 Years
R0 Resection Rate | 6 Month
Treatment RelatedToxicity | 3 Year
  Adverse events grade that greater than 3 is considered secondary endpoint, according to the Common Terminology Criteria for Adverse Events Version 3.0.
Life Quality | 3 Years
  EORTC QoL Questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Ping Lan, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The 6th Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China